CLINICAL TRIAL: NCT03722758
Title: Clinical Performance of a Micro-hybride Resin Based Composite in the Treatment of Cervical Caries Lesions: 36-month, Split-mouth, Randomized Clinical Trial
Brief Title: 36-Month Clinical Performance of Different Restorative Materials in the Treatment of Root Caries Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Uzay Koc, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2016/03-23 (KA-16003)
Record Dates: First submitted 2018-10-24; First posted 2018-10-29 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Root Caries
Keywords: micro hybrid resin composite; resin-modified glass ionomer; split-mouth randomized clinical trial
MeSH Terms: conditions — Root Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spectrum TPH3, tooth restoration (Active Comparator): Restoration with micro hybrid resin composite
  Interventions: Device: Spectrum TPH3; Device: Riva LC
- Riva LC, restorative material (Active Comparator): Restoration with resin-modified glass ionomer cement
  Interventions: Device: Spectrum TPH3; Device: Riva LC

INTERVENTIONS:
Device: Spectrum TPH3 — tooth restoration with two different restorative materials
  Other Names: resin composite
Device: Riva LC — tooth restoration with two different restorative materials
  Other Names: RMGİC

SUMMARY:
This is a split-mouth, randomized clinical study that evaluating the 36-month performance of different restorative materials in the treatment of root caries lesions. A total of 110 restorations were randomly placed, half using resin composite (Spectrum TPH3) and the other half using the resin-modified glass ionomer cement (Riva Light Cure). Restorations were evaluated at the baseline, 6, 12, 18,24 and 36 months according to the USPHS criteria.

DETAILED DESCRIPTION:
The aim of the study was to comparatively assess the 36-month clinical performance of a micro hybrid resin composite and resin-modified glass ionomer cement in root caries lesions.

Thirty-three patients with at least two root caries lesions participated in this study. A total of 110 restorations were randomly placed, half using resin composite (Spectrum TPH3) and the other half using the resin-modified glass ionomer cement (Riva Light Cure). Restorations were evaluated at the baseline, 6, 12, 18, 24 and 36 months. The data were analyzed with Pearson's Chi-square, Cochran's Q, Friedman tests and Logistic Regression Analysis (p=0.05).

ELIGIBILITY:
Inclusion Criteria:

* Root caries lesions (at least 1mm depth)

Exclusion Criteria:

* Complex medical history
* Poor dental hygiene/infrequent practise of oral hygiene habits
* Severe or chronic periodontitis
* Extreme carious activity
* Heavy bruxism
* Very deep (closer than 0.5 mm to the pulp) or superficial lesions (shallower than 1mm)
* Previously restored and abutment teeth for bridge or removable dental prostheses

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-07-15 (Actual); Primary Completion 2018-07-15 (Actual); Study Completion 2019-11-15 (Estimated)

PRIMARY OUTCOMES:
Marginal adaptation 0 for at least 90% restorations (marginal adaption score) | 24 months
  The primary factor for determining the clinical performance of a restorative material is the marginal adaption score. It represents the survival rates of the restorations after a period of time. According to ADA guidelines, a restorative material should show at least 90% survival rate after 18. The retention scored as 0 (restoration appears to adapt closely to the surface of the tooth with no crevice formation), 1 (an explorer caught lightly when run in both directions, and there was visible evidence of early crevice formation), 2 (an explorer got caught in both directions and penetrated a marginal crevice), 3 (the crevice had sufficient depth to expose the dentin, required replacement) or 4 (The restoration was fractured or lost).
  Clinical evaluation is performed to examine if the restorations are in place or fallen.

CONTACTS AND LOCATIONS:
Overall Officials: Uzay Koc-Vural, Principal Investigator — Hacettepe University